CLINICAL TRIAL: NCT00006108
Title: A Phase II Trial of Xeloda, Every Three Week Taxol and Herceptin in Metastatic Breast Cancer
Brief Title: Capecitabine, Paclitaxel, and Trastuzumab in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: LCCC 9904; UNC-9904; NCI-G00-1834 (Registry Identifier: National Cancer Institute); CDR0000068119 (Other: PDQ number)
Record Dates: First submitted 2000-08-03; First posted 2004-02-26 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Capecitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: trastuzumab
Drug: capecitabine
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining chemotherapy with monoclonal antibody therapy may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining capecitabine, paclitaxel, and trastuzumab in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of capecitabine when administered in combination with paclitaxel and trastuzumab (Herceptin) in patients with metastatic breast cancer. II. Determine the response rate of these patients to this treatment regimen. III. Determine the median time to treatment failure in these patients with this treatment regimen. IV. Determine the incidence of cardiac toxicity in these patients with this treatment regimen. V. Assess the quality of life in these patients.

OUTLINE: This is a dose escalation study of capecitabine. Patients receive trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15; paclitaxel IV over 3 hours on day 2; and oral capecitabine on days 3-16. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Once the MTD is determined, additional patients are accrued. Quality of life is assessed at baseline and after 3 courses of treatment.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for the phase I dose escalation portion of this study. A total of 28-41 patients will be accrued for the phase II portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the breast Metastatic disease HER2 overexpressing tumor (2+ or 3+) Bidimensionally measurable or evaluable disease Hormone receptor status: Estrogen receptor positive or negative

PATIENT CHARACTERISTICS: Age: 18 to 59 Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal Renal: Creatinine less than 1.5 mg/dL Cardiovascular: Ejection fraction at least 50% by MUGA No history of congestive heart failure No uncontrolled cardiac arrhythmias Other: No other prior malignancy except squamous cell or basal cell carcinoma of the skin, noninvasive ductal carcinoma of the breast, or cervical dysplasia No prior motor or sensory neuropathy grade 2 or higher Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior trastuzumab (Herceptin) No concurrent hematopoietic growth factors Chemotherapy: No prior chemotherapy for metastatic disease Prior adjuvant chemotherapy allowed (including regimens containing doxorubicin) No prior paclitaxel, 24 hour infusion fluorouracil, or capecitabine Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to 50% or more of the bone marrow Surgery: Not specified Other: No other concurrent experimental drugs

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1999-08; Primary Completion 2001-09 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances A. Collichio, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina, United States